CLINICAL TRIAL: NCT05541757
Title: In-Vitro Evaluation of Anticoagulant Therapy Management When Urgent Percutaneous Coronary Intervention is Required in Rivaroxaban-Treated Patients
Brief Title: Rivaroxaban - Percutaneous Coronary Intervention
Status: Completed | Type: Observational
Sponsor: Bursa Postgraduate Hospital (Other)
Responsible Party: Principal Investigator, Hasan ARI, Professor Doctor, Bursa Postgraduate Hospital
Other Study IDs: BYİEAH4
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Coronary Artery Disease; Atrial Fibrillation
MeSH Terms: conditions — Coronary Artery Disease; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: five healthy adults
  Interventions: Drug: In vitro heparin
- Study group: Twenty-five patients using the direct oral factor Xa inhibitor rivaroxaban
  Interventions: Drug: In vitro heparin

INTERVENTIONS:
Drug: In vitro heparin — In vitro heparin and in vitro LMWH

SUMMARY:
We investigated in-vitro the management of intraprocedural anticoagulation in patients requiring immediate percutaneous coronary intervention(PCI) while using regular direct oral anticoagulants(DOACs). Twenty-five patients taking 20mg of rivaroxaban once daily comprised the study group, while five healthy volunteers included the control group. In study group, a beginning(24-hours after the last rivaroxaban dose) examination was performed. Then, the effects of basal and four different anticoagulant doses(50IU/kg unfractionated heparin(UFH), 100IU/kg UFH, 0.5mg/kg enoxaparin, and 1mg/kg enoxaparin) on coagulation parameters were investigated at the 4th and 12th hours following rivaroxaban intake. Anticoagulant activity was assessed mainly by anti-factor Xa(anti-Xa) levels.

ELIGIBILITY:
Inclusion Criteria:

* patients using the direct oral factor Xa inhibitor rivaroxaban
* Atrial fibrillation

Exclusion Criteria:

* malignancy,
* coagulopathy,
* heart valve disease,
* active infection,
* chronic systemic or inflammatory disease,
* recent ACS or elective PCI,
* uncontrolled hypertension and diabetes,
* cerebrovascular accident,
* thyroid disorder,
* left ventricular systolic dysfunction (ejection fraction <50%),
* glomerular filtration rate <50 mL/min/1.73 m2,
* underweight and overweight (<60 kg and >100 kg),
* age >75 years,
* hyperbilirubinemia and hypertriglyceridemia (>350 mg/dl).

Ages: 18 Years to 74 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with persistent or permanent AF had been using rivaroxaban 20 mg daily for at least one month
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Anticoagulation level | 4 - 12 hours
  anti-factor Xa

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yüksek İhtisas Eğitim ve Araştırma Hastanesi, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Melek M, Ari H, Ari S, Cilgin MC, Yarar M, Huysal K, Agca FV, Bozat T. In vitro evaluation of anticoagulant therapy management when urgent percutaneous coronary intervention is required in rivaroxaban-treated patients. Naunyn Schmiedebergs Arch Pharmacol. 2023 Nov;396(11):3221-3232. doi: 10.1007/s00210-023-02533-2. Epub 2023 May 20. PMID 37209152